CLINICAL TRIAL: NCT06535269
Title: Prospective Randomized Study on Postoperative Pain in the Surgical Treatment of Hemorrhoids Through Conventional Hemorrhoidectomy With a Monopolar Electric Scalpel or Bipolar Energy With Caiman® (Aesculap®)
Brief Title: Postoperative Pain in the Surgical Treatment of Hemorrhoids: Conventional Hemorrhoidectomy With a Monopolar Electric Scaler VS Bipolar Energy With Caiman® (Aesculap®)
Acronym: TAUHEMOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Laura Mora-Lopez, PhD, MD, Colorrectal Surgeon, Associate Professor, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAUHEMOR
Record Dates: First submitted 2024-07-11; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Hemorrhoid Pain; Hemorrhoidectomy

STUDY DESIGN:
Intervention Model Description: Non-inferiority, prospective, randomized, single-center, parallel-group clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Conventional hemorrhoidectomy with monopolar diathermy + intravenous analgesia with elastomeric pump + discharge with home hospitalization.
  Interventions: Procedure: Monopolar Hemorroidecotmy
- Experimental (Experimental): conventional haemorrhoidectomy with Caiman® bipolar energy (AESCULAP®) + oral conventional analgesia + conventional home discharge.
  Interventions: Procedure: Caiman Hemorroidectomy

INTERVENTIONS:
Procedure: Monopolar Hemorroidecotmy — Hemorrhoidectomy with monopolar diathermy
  Arms: Control
Procedure: Caiman Hemorroidectomy — Hemorrhoidectomy with Caiman® bipolar energy
  Arms: Experimental

SUMMARY:
To demonstrate that postoperative pain secondary to Milligan and Morgan hemorrhoidectomy with Caiman® (AESCULAP®) and subsequent oral conventional analgesia is at least not greater than that generated after hemorrhoidectomy with monopolar diathermy and intravenous analgesia with care home at discharge.

DETAILED DESCRIPTION:
In the treatment of coloproctological pathology, one of the most important problems is postoperative pain. Especially in the management of hemorrhoids treatment. There are different approaches but in all of them pain is the predominant symptom.

There are some less painful techniques but the gold standard continues to be hemmorrhoidectomy, which is associated with postoperative pain. Some actions have been taken to control pain to avoid the admission of patients, but there are still problems in this regard.

Our group aims to study the effect of energy change for performing hemorrhoidectomy on postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* All patients with 2 or 3 bundles of grade III-IV hemorrhoids (Goligher classification) clinically symptomatic and subject to outpatient hemorrhoidectomy
* Voluntary participation.
* ASA I-II-III.

Exclusion Criteria:

* Failure to meet the inclusion criteria.
* ASA IV.
* Allergic to Paracetamol, derivatives of morphine.
* Allergic to NSAIDs.
* Synchronous colorectal neoplasia.
* Coagulation disorders.
* Thrombosed hemorrhoid.
* Inflammatory bowel disease.
* Liver cirrhosis and/or portal hypertension.
* Pregnant women.
* Difficulty following up by phone and/or in person.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 6 hours of post-operative period (before hospital discharge performed); within 2 days with telephone control; at 7 days control at external consultations; at 30 days control at external consultations
  Postoperative pain: value 0 (no pain) - 10 (maximum pain)

SECONDARY OUTCOMES:
Wound healing time | 7 days postoperative control at external consultations; 30 days postoperative control at external consultations
  A healed wound is considered when all post-hemorrhoidectomy wounds of 2-3 bundles are epithelialized
Post-surgery satisfaction survey | 30 days postoperative control at external consultations
  Phone checklist survey
Wexner scale | in pre-operative visit, on the 7th and 30th postoperative clinical control
  Assessment of fecal incontinence o a scale from 0 (never incontinence) to 4 (always), obtaining a score between 0 and 20.
Number of emergency consultations | in 30 days post-surgery
  revision of Database
Collection of adverse effects from patients | in 30 days post-surgery
  revision of Database

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mora, Principal Investigator — Parc Tauli University Hospital
Locations (1):
- Laura Mora López, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perera N, Liolitsa D, Iype S, Croxford A, Yassin M, Lang P, Ukaegbu O, van Issum C. Phlebotonics for haemorrhoids. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD004322. doi: 10.1002/14651858.CD004322.pub3. PMID 22895941
- [Background] Alonso-Coello P, Guyatt G, Heels-Ansdell D, Johanson JF, Lopez-Yarto M, Mills E, Zhou Q. Laxatives for the treatment of hemorrhoids. Cochrane Database Syst Rev. 2005 Oct 19;2005(4):CD004649. doi: 10.1002/14651858.CD004649.pub2. PMID 16235372
- [Background] Shanmugam V, Thaha MA, Rabindranath KS, Campbell KL, Steele RJ, Loudon MA. Rubber band ligation versus excisional haemorrhoidectomy for haemorrhoids. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD005034. doi: 10.1002/14651858.CD005034.pub2. PMID 16034963
- [Background] Medina-Gallardo A, Curbelo-Pena Y, De Castro X, Roura-Poch P, Roca-Closa J, De Caralt-Mestres E. Is the severe pain after Milligan-Morgan hemorrhoidectomy still currently remaining a major postoperative problem despite being one of the oldest surgical techniques described? A case series of 117 consecutive patients. Int J Surg Case Rep. 2017;30:73-75. doi: 10.1016/j.ijscr.2016.11.018. Epub 2016 Nov 15. PMID 27960130
- [Background] Nienhuijs S, de Hingh I. Conventional versus LigaSure hemorrhoidectomy for patients with symptomatic Hemorrhoids. Cochrane Database Syst Rev. 2009 Jan 21;2009(1):CD006761. doi: 10.1002/14651858.CD006761.pub2. PMID 19160300
- [Background] Gentile M, De Rosa M, Carbone G, Pilone V, Mosella F, Forestieri P. LigaSure Haemorrhoidectomy versus Conventional Diathermy for IV-Degree Haemorrhoids: Is It the Treatment of Choice? A Randomized, Clinical Trial. ISRN Gastroenterol. 2011;2011:467258. doi: 10.5402/2011/467258. Epub 2010 Nov 21. PMID 21991510
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krle A-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 Statement: defining standard protocol items for clinical trials. Rev Panam Salud Publica. 2015 Dec;38(6):506-14. PMID 27440100